CLINICAL TRIAL: NCT07067632
Title: Mortality Outcome of Controlled Hypertension in Randomized Controlled or Open-label Study Intentionally Directed Intervention Effect Blood Pressure: A Systematic Review and Meta-Analysis
Brief Title: To Study the Mortality Outcome of Controlled Blood Pressure Participants
Acronym: HTN-Mort
Status: Recruiting | Type: Observational
Sponsor: DejthidaNathaphong (Other)
Responsible Party: Sponsor
Other Study IDs: DejthidaNathaphong
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Valid MeSH Conditions; Hypertension (HTN)
Keywords: hypertension; cardiovascular death
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antihypertensive treatment: Participants assigned to interventions (pharmacological, device-based, or lifestyle) directed at lowering blood pressure or Antihypertensive agents, Blood pressure-lowering treatment, Antihypertensive therapy.
  Interventions: Drug: Antihypertensive treatment
- Control/Comparator: Participants receiving placebo, standard of care, or no intervention

INTERVENTIONS:
Drug: Antihypertensive treatment — Any intervention (pharmacological, device-based, lifestyle) intentionally directed at lowering BP
  Control groups receiving placebo, standard of care, or no intervention
  Other Names: device-based blood pressure lowering; lifestyle modification
  Groups: Antihypertensive treatment

SUMMARY:
Despite advances in antihypertensive therapy, some patients with well-controlled blood pressure still experience fatal outcomes. This paradox raises critical questions about the efficacy of blood pressure-targeted interventions and whether BP control alone ensures survival. This systematic review and meta-analysis aims to evaluate all-cause mortality and cardiovascular death among hypertensive patients who achieved BP targets in RCTs or open-label trials.

To determine whether achieving controlled blood pressure through intentional intervention (pharmacological or procedural) in RCTs or open-label studies reduces mortality (all-cause and cardiovascular) in hypertensive patients.

DETAILED DESCRIPTION:
Sensitivity Analyses Excluding high risk of bias studies

Excluding short follow-up (<1 year)

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with diagnosed hypertension

Blood pressure controlled at target values defined by the study (e.g., <140/90 mmHg or <130/80 mmHg)

Any comorbidity allowed unless the study focuses on pregnancy or pediatric population

Exclusion Criteria:

* Observational or retrospective studies

Pediatric or pregnant participants

Case reports, editorials, or conference abstracts without full data

Studies not reporting mortality outcomes separately for controlled BP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥18 years with diagnosed hypertension
  Blood pressure controlled at target values defined by the study (e.g., <140/90 mmHg or <130/80 mmHg)
  Any comorbidity allowed unless the study focuses on pregnancy or pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 100 year
  All cause mortality by controlable hypertension treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nathaphong Dejthida, MD, Principal Investigator — DejthidaNathaphong
Locations (1):
- Nathaphong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No